CLINICAL TRIAL: NCT02954575
Title: Clinical Study to Investigate the Pharmacokinetics, Efficacy, Safety, and Immunogenicity of Wilate in Previously Treated Patients With Severe Hemophilia A
Brief Title: Clinical Study to Investigate the PK, Efficacy, and Safety of Wilate in Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIL-27
Record Dates: First submitted 2016-10-27; First posted 2016-11-03 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — von Willebrand Factor; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients will receive Wilate for prophylactic treatment
  Interventions: Drug: Wilate

INTERVENTIONS:
Drug: Wilate
  Other Names: von Willebrand factor / Factor VIII (plasma derived)

SUMMARY:
The purpose of this study is to obtain additional data on the safety and efficacy of Wilate in PTPs with hemophilia A with at least 150 previous exposure days (EDs) to a FVIII concentrate who undergo prophylactic treatment with Wilate for 6 months and at least 50 EDs, thus supplementing the existing database to obtain approval of Wilate for the indication hemophilia A in the USA.

ELIGIBILITY:
Inclusion Criteria:

1. Severe hemophilia A (<1% FVIII:C) according to medical history
2. Male patients aged ≥12 years
3. Previous treatment with a FVIII concentrate for at least 150 exposure days (EDs)
4. Immunocompetence (CD4+ count >200/µL)
5. Good documentation of the historical bleeding rate (at least for the 6 months preceding study start)
6. Voluntarily given, fully informed written and signed consent obtained by the patient (or parent/legal guardian in case of adolescents) before any study-related procedures are conducted

Whenever possible, the interval between the Screening Visit and the PK or Non-PK Visit should not exceed 30 days. If the 30-day interval is exceeded, determination of the CD4+ count is to be repeated and must be >200/µL for patients to be enrolled (i.e., exclusion criterion no. 4).

Exclusion Criteria:

1. Any coagulation disorders other than hemophilia A
2. History of FVIII inhibitor activity (≥0.6 BU) or detectable FVIII inhibitory anti-bodies (≥0.6 BU using the Nijmegen modification of the Bethesda assay) at screening, as determined by the central laboratory
3. Severe liver or kidney diseases (alanine aminotransferase [ALAT] and aspartate transaminase [ASAT] levels >5 times of upper limit of normal, creatinine>120 µmol/L)
4. Patients receiving or scheduled to receive immunomodulating drugs (other than anti-retroviral chemotherapy) such as alpha-interferon, prednisone (equivalent to >10 mg/day), or similar drugs
5. Treatment with any investigational medicinal product in another interventional clinical study currently or within 4 weeks before enrollment

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Solomon, MD, Study Director — Octapharma
Locations (7):
- Specialized Hospital for Active Treatment "Joan Pavel", Sofia, Bulgaria
- National Haemophilia Centre, Budapest, Hungary
- Poland (2):
  - Krakowskie Centrum Medyczne, Krakow
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
- Centrul Medical Unirea -Policlinica Enescu, Bucharest, Romania
- Russia (2):
  - Barnaul Branch of RAMS hematology center, Barnaul
  - Federal Scientific Hematology Center, Moscow

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wilate: A total of 57 patients were enrolled in the study. For the PK assessment (PK population) a single dose of Wilate of 50 ±5 IU/kg BW was administered to 21 patients.
  For prophylactic treatment, Wilate was administered every 2 to 3 days at a dose of 20-40 IU/kg BW for 6 months. In case of unacceptably frequent spontaneous breakthrough BEs, the dose of Wilate was increased by approximately 5 IU/kg.
  The dose (and duration) of treatment for BEs was dependent on the location and extent of bleeding and on the clinical condition of the patient; range: 10-50 IU/kg every 12-24 hours or 8-24 hours until resolved.
  For the surgical prophylaxis population (SURG population), minor surgeries were treated with 15-30 IU/kg every 24 hours, at least 1 day, until healing iwas achieved. Major surgeries were treated with 40-50 IU/kg, repeat injection every 8-24 hours until adequate wound healing, then therapy for at least another 7 days to maintain a FVIII activity of 30% to 60%.
Period: Overall Study
Arm/Group | Wilate
Started | 57
Received Treatment | 55
SAF Population (SAF population = study population of patients in safety analysis) | 55
FAS Population (FAS population = full analysis population) | 55
PP Population (PP population = per-protocol population) | 52
PK Population (PK population = study population of patients who underwent pharmacokinetic analysis) | 21
SURG Population (SURG population = study population of patients undergoing surgery treated with Wilate) | 1
Completed | 54
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The safety (SAF) population includes all patients who received at least one administration of Wilate during the study (N=55)
Groups:
- Wilate: SAF population (All patients who received at least one administration of Wilate during the study (N=55)
Arm/Group | Wilate
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 83.3 (21.4)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 26.8 (5.8)
Blood groups [Count of Participants; unit: Participants]
  0 | 19
  A | 23
  AB | 5
  B | 8
von Willebrand factor antigen (VWF:Ag) [Mean (Standard Deviation); unit: IU/dL] — Plasma VWF:Ag measurements recorded at baseline
  IU/dL | 118.4 (78.9)
von Willebrand factor activity (VWF:Ac) [Mean (Standard Deviation); unit: IU/dL] — Plasma VWF:Ac measurements recorded at baseline
  IU/dL | 103.7 (39.5)
Previous Factor (F) VIII treatment [Count of Participants; unit: Participants]
  On-demand | 32
  Prophylaxis | 18
  Combination | 5
Previous annualized bleeding rate (ABR) [Mean (Standard Deviation); unit: No. BEs per patient per year] — Previous ABR is based on the bleeding rate in the 6 months prior to entry into the study.
  No. BEs per patient per year | 32.98 (39.12)

OUTCOME MEASURES:

1. Primary Outcome: Total Annualized Bleeding Rate (TABR)
Description: The total number of bleeding events (BEs) was documented by patients in a patient diary (together with the investigator in case of on-site treatments), which was reviewed at each follow-up visit by site personnel.
Time Frame: 6 months
Population: The total annualized bleeding rate (TABR) was calculated for all patients included in the PP population (N=52).
Measure: Mean (Standard Deviation); unit: No. of BEs / year (ABR)
Units Other Than Participants: No. of Bleeding Episodes (BEs)
Groups:
- Wilate: PP population
Arm/Group | Wilate
Number analyzed (Participants) | 52
Number analyzed (No. of Bleeding Episodes (BEs)) | 57
No. of BEs / year (ABR) | 2.10 (3.44)
Statistical Analysis 1: Comparison: Wilate; A confirmative one-sided, one-sample Poisson test was used to test whether the mean annualized bleeding rate (ABR) in patients treated prophylactically with Wilate was below the threshold of 29 BEs per patient year (alpha = 2.5%). This threshold corresponds to 50% of the TABR reported in the GENA-01 study (NCT00989196), which observed 58.1 BEs per patient per year. A corresponding two-sided 95% CI for the TABR was also analyzed; Test type: Other; p < 0.0001, Poisson test estimate — versus mean TABR >29; Poisson test estimate = 2.13, 95% CI 2-sided [1.64 to 2.76]

2. Secondary Outcome: Spontaneous Annualized Bleeding Rate (SABR)
Description: The number of spontaneous bleeding events (BEs) was documented by patients in a patient diary (together with the investigator in case of on-site treatments), which was reviewed at each follow-up visit by site personnel.
Time Frame: 6 months
Population: The spontaneous annualized bleeding rate (SABR) was calculated for all patients included in the PP population (N=52).
Measure: Mean (Standard Deviation); unit: No. of spontaneous BEs/year (SABR)
Units Other Than Participants: No. of BEs
Arm/Group | Wilate
Number analyzed (Participants) | 52
Number analyzed (No. of BEs) | 41
No. of spontaneous BEs/year (SABR) | 1.51 (3.03)
Statistical Analysis 1: Comparison: Wilate; A confirmative one-sided, one-sample Poisson test was used to test whether the mean SABR in patients treated prophylactically with Wilate was below the threshold of 19.1 BEs per patient year (alpha = 2.5%). This threshold corresponds to 50% of the SABR in the GENA-01 study (NCT00989196), which observed 38.2 spontaneous BEs per patient per year. A corresponding two-sided 95% CI for the SABR was also analyzed; Test type: Other; p < 0.0001, Poisson test estimate — versus mean SABR >19.1; Poisson test estimate = 1.53, 95% CI 2-sided [1.13 to 2.08]

3. Secondary Outcome: Efficacy of Wilate in the Treatment of Breakthrough BEs
Description: The proportion of BEs successfully treated with Wilate were documented by the patient (together with the investigator in case of on-site treatments) in the patient diary for all BEs according to a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none', where 'excellent' was defined as "Abrupt pain relief and/or unequivocal improvement in objective signs of bleeding within approximately 8 hours after a single injection" (best outcome) and 'none' was defined as "No improvement within 12 hours, or worsening of symptoms, requiring more than two injections for complete resolution" (worst outcome). All efficacy ratings assessed as either 'excellent' or 'good' were considered 'successfully treated.'
Time Frame: 6 months
Population: In the PP population, efficacy of Wilate in the treatment of breakthrough BEs was analyzed for all patients experiencing breakthrough BEs (N=24)
Measure: Count of Units; unit: Number of BEs
Units Other Than Participants: Number of BEs
Groups:
- Wilate: Efficacy of Wilate was analysed for the PP population
Arm/Group | Wilate
Number analyzed (Participants) | 24
Number analyzed (Number of BEs) | 57
Number of BEs
  Excellent | 16
  Good | 32
  Moderate | 9
Statistical Analysis 1: Comparison: Wilate; Confirmatory statistical testing tested the null hypotheses that the percentage of success is ≤70% (alternative hypothesis: percentage >70%); the test procedure based on the generalized estimation equation took into account several BEs in one patient as correlated repeated measurements (alpha = 2.5%). Thus, π denotes the proportion of success and the following pair of hypotheses was tested: H0: π ≤ 0.7 vs. H1: π > 0.7; Test type: Other; p = 0.0096, Confirmatory data analysis; Generalized estimation equation = 84.21, 95% CI 2-sided [72.13 to 92.52]

4. Secondary Outcome: Wilate Consumption Data (Average Total Normdose of FVIII IU/kg Per Month of Study) for Prophylaxis
Description: The average consumption of Wilate per month of study (IU/kg) for all patients receiving prophylaxis.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Wilate
Number analyzed (Participants) | 52
IU/kg | 405.06 (83.70)

5. Secondary Outcome: Pharmacokinetic (PK) Assessment (Area Under the Curve [AUC] Norm) of FVIII:C
Description: PK assessments of FVIII:C were conducted using the one-stage (OS) assay. The value of the AUCnorm of FVIII:C was calculated based on the FVIII:C values measured in the patients participating in the PK study.
Time Frame: Initial PK visit (Day -1) and PK study completion visit (6 months); data collected 1 h prior to injection and 15 min, 1 h, 3 h, 6 h, 9 h, 24 h, 30 h and 48 h after the end of injection
Population: AUC divided by dose (IU*h/dL per IU/kg)
Measure: Mean (Standard Deviation); unit: IU*h/dL per IU/kg
Groups:
- Wilate: PK population
Arm/Group | Wilate
Number analyzed (Participants) | 21
IU*h/dL per IU/kg
  Initial PK | 28.61 (9.31)
  PK completion 6 months | 30.75 (11.32)

6. Secondary Outcome: Pharmacokinetic (PK) Assessment (in Vivo Half-Life (t1/2)) of FVIII:C
Description: PK assessments of FVIII:C were conducted using the one-stage (OS) assay. The in vivo half-life of FVIII:C was calculated based on the FVIII:C values measured in the patients participating in the PK study.
Time Frame: Initial PK assessment (Day -1) and PK study completion visit (6 months); data collected 1 h prior to infusion and 15 min, 1 h, 3 h, 6 h, 9 h, 24 h, 30 h and 48 h after the end of injection
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Wilate
Number analyzed (Participants) | 21
Hours
  Initial PK | 10.82 (2.50)
  PK completion 6 months | 11.50 (2.30)

7. Secondary Outcome: Pharmacokinetic (PK) Assessment (Maximum Plasma Concentration [Cmax]) of FVIII:C
Description: PK assessments of FVIII:C were conducted using the one-stage (OS) assay. The maximum plasma concentration of FVIII:C was calculated based on the FVIII:C values measured in the patients participating in the PK study.
Time Frame: Initial PK assessment (Day -1) and 6 months
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Wilate
Number analyzed (Participants) | 21
IU/dL
  Initial PK | 106.70 (22.45)
  PK completion 6 months | 103.49 (26.53)

8. Secondary Outcome: Incremental in Vivo Recovery (IVR) of Wilate Over Time
Description: The rise in FVIII activity in IU/dl per unit dose administered in IU/kg was determined from all patients at baseline, 3 and 6 months, using the OS assay.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: kg/dL
Groups:
- Wilate: FAS population
Arm/Group | Wilate
Number analyzed (Participants) | 55
kg/dL
  First PK/non-PK visit | 2.14 (0.51)
  3 months | 2.14 (0.49)
  PK/non-PK completion 6 months | 1.97 (0.64)

9. Secondary Outcome: Association Between ABO Blood Type and the FVIII:C Half-life of Wilate (OS Assay)
Description: Analysis of variance (ANOVA) was used in an exploratory sense to assess an association between ABO blood type and the FVIII:C half-life of Wilate. This was analyzed by calculating the mean square in a one-stage assay.
Time Frame: 6 months
Measure: Number; unit: Beta coefficient
Arm/Group | Wilate
Number analyzed (Participants) | 21
Beta coefficient | 15.867
Statistical Analysis 1: Comparison: Wilate; Test type: Other; p = 0.0346, ANOVA

10. Secondary Outcome: Association Between VWF:Ag Concentration and the FVIII:C Half-life of Wilate
Description: ANOVA was used in an exploratory sense to assess an association between VWF:Ag with the FVIII:C half-life of Wilate. This was analyzed by calculating the mean square in a one-stage assay.
Time Frame: 6 months
Measure: Number; unit: Beta coefficient
Arm/Group | Wilate
Number analyzed (Participants) | 21
Beta coefficient | 5.104
Statistical Analysis 1: Comparison: Wilate; Test type: Other; p = 0.4244, ANOVA

11. Secondary Outcome: Safety and Tolerability of Wilate by Monitoring Adverse Events (AEs) Throughout the Study
Description: At each (scheduled or unscheduled) study visit, AEs were documented by the investigator throughout the study.
Time Frame: 6 months
Population: In the FAS population (N=55), the safety and tolerability of Wilate was analysed for all patients experiencing adverse events (AEs) throughout the study.
Measure: Number; unit: Number of adverse events
Arm/Group | Wilate
Number analyzed (Participants) | 55
Number of adverse events
  Number of AEs | 17
  Number of Treatment-emergent AEs | 16

12. Secondary Outcome: Immunogenicity of Wilate by Testing for FVIII Inhibitors
Description: FVIII inhibitor activity was determined at each study visit before the injection of Wilate using the modified Bethesda assay (Nijmegen modification).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Wilate
Number analyzed (Participants) | 55
Participants | 0
Statistical Analysis 1: Comparison: Wilate; Test type: Other; Pearson-Copper = 0, 95% CI 2-sided [0 to 16.11]

13. Secondary Outcome: Virus Safety Measured by the Number of Parvovirus B19 Seroconversions Between Baseline (BL) and End of Study
Description: Virus safety was evaluated by taking a plasma sample for parvovirus B19 antibody testing before the first injection of Wilate. All patients negative at screening were tested again at the study completion visit. The number with Parvovirus B19 seroconversions between BL and end of study was recorded.
Time Frame: 6 months
Population: In the FAS population (N=55), the viral safety of Wilate was analyzed for all patients at baseline.
Measure: Number; unit: Participants
Arm/Group | Wilate
Number analyzed (Participants) | 55
Participants | 0

14. Other Pre Specified Outcome: Efficacy of Wilate in Surgical Prophylaxis
Description: Hemostatic efficacy was assessed at the end of surgery by the surgeon and at end of the postoperative period by the hematologist, using a 4-point hemostatic efficacy scale including the four items: 'excellent' (best possible outcome), 'good', 'moderate' and 'none' (worst outcome). Overall efficacy was assessed by the investigator, taking both the intra and postoperative assessments into account, and using the 'excellent,' 'good,' moderate,' and 'none' scale.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Wilate: SURG population (study population of patients undergoing surgery treated with Wilate)
Arm/Group | Wilate
Number analyzed (Participants) | 1
Participants
  Excellent | 0
  Good | 1
  Moderate | 0
  None | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Wilate: SAF population
Arm/Group | Wilate
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 12/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wilate (N=55)
Erysipelas (Infections and infestations) | 1 (1) — Treatment-emergent adverse event
Nasopharyngitis (Infections and infestations) | 1 (1) — Treatment-emergent adverse event
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) — Treatment-emergent adverse event
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) — Treatment-emergent adverse event
Seasonal allergy (Immune system disorders) | 2 (2) — Treatment-emergent adverse event
Headache (Nervous system disorders) | 1 (1) — Treatment-emergent adverse event
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) — Treatment-emergent adverse event
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5) — Treatment-emergent adverse event
Pain (General disorders) | 1 (1) — Treatment-emergent adverse event
Limb injury (Injury, poisoning and procedural complications) | 1 (1) — Treatment-emergent adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT02954575/Prot_002.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02954575/SAP_003.pdf